CLINICAL TRIAL: NCT01815086
Title: Radioimmunoimaging (PET/CT) of Patients With AL Amyloidosis Using the 124I-Labeled Amyloid-Reactive Monoclonal Antibody (mAb) Murine (Mu) 11-F4
Brief Title: Radioimmunoimaging of Light Chain (AL) Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Alan Solomon, Professor of Mediciine; Head, Human Immunology & Cancer Program, FDA Office of Orphan Products Development
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IND 100472; 1R01FD003420-01A1 (FDA)
Record Dates: First submitted 2013-03-13; First posted 2013-03-20 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: AL Amyloidosis
Keywords: Radioimmunoimaging; AL Amyloidosis; PET/CT
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 124I-labeled anti-amyloid mAb 11-1F4 (Experimental): 124I-labeled anti-amyloid mAb 11-1F4 will be infused on day 0. Two and 5 days later, PET/CT scans will be performed.
  Interventions: Biological: Single infusion of 124I-labeled anti-amyloid mAb 11-1F4: 2 mCi (1 mg)

INTERVENTIONS:
Biological: Single infusion of 124I-labeled anti-amyloid mAb 11-1F4: 2 mCi (1 mg) — Single infusion of 124I-labeled anti-amyloid mAb 11-1F4: 2 mCi (1 mg)

SUMMARY:
The purpose of the study is to determine the capability of a radiolabeled amyloid-reactive monoclonal antibody (mAb) to document the presence and distribution of amyloid deposits by PET/CT imaging in patients with AL amyloidosis.

DETAILED DESCRIPTION:
To be eligible for this study, patients must have a confirmed diagnosis of AL amyloidosis without significant cardiac (New York Heart Association class IV) disease and not be on kidney dialysis. Additionally, after testing, their blood must not contain antibodies to mouse proteins. The study requires an intravenous infusion, given over 10 minutes, of the radiolabeled antibody, followed 48 hours later by a PET/CT scan. A repeat scan is done 5 days after infusion of the antibody. A 5-ml blood specimen needs to be furnished 4 and 8 weeks after the antibody infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of AL amyloidosis.

Exclusion Criteria:

* New York Heart Association class IV
* On renal dialysis
* Serum antibodies to mouse protein

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determination of the capability of a radiolabeled amyloid-reactive monoclonal antibody (mAb) to document the presence and distribution of amyloid deposits by PET/CT in up to 30 patients with AL amyloidosis. | Five days post PET/CT scan
  PET/CT images will be taken 2 and 5 days post-radiolabeled antibody infusion to evaluate if there is organ/tissue uptake (greater than blood pool) and to determine if the presence of radiolabeled antibody correlates with clinically proven amyloid deposition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States